CLINICAL TRIAL: NCT05211531
Title: Walk With a Doc: Enhanced Recovery Walking Program for Surgical Inpatients and Wellness Program for Surgical Residents
Acronym: WWAD
Status: Terminated | Type: Observational
Why Stopped: Lead study team member deceased, project not continued.
Sponsor: Richard Perugini (Other)
Collaborators: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor-Investigator, Richard Perugini, Assistant Professor, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Other Study IDs: H00019609
Record Dates: First submitted 2022-01-11; First posted 2022-01-27 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Complication of Surgical Procedure; Resident Physicians
Keywords: Resident physician wellness; Post-operative walking program

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measuring number of post-operative steps — Measuring the number of post-operative steps that inpatients take.

SUMMARY:
Program studying the number of steps post-operative patients need to take to prevent post-operative complications. Also studying surgical resident wellness program that provides extra time to ambulate with inpatients.

DETAILED DESCRIPTION:
Program studying the number of steps post-operative patients need to take to prevent post-operative complications. Patients receive a pedometer while inpatient to measure their daily steps, which is recorded in the electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

* Post-operative surgical patient with an over 24 hour post-operative stay in the hospital
* Safe to ambulate with/without assistance

Exclusion Criteria:

* Unable to ambulate
* Bedbound

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Minimally invasive surgery patients who are admitted and undergo surgery at a single tertiary care center.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Total number of steps | From index surgery to initial post-operative office visit, up to 3 weeks
  Total number of steps ambulated by the patient as measured by a pedometer
30 day Post-operative complications | 30 days
  30 day Post-operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Richard Perugini, MD, Principal Investigator — UMASS Memorial Healthcare
Locations (1):
- UMASS Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No